CLINICAL TRIAL: NCT01865812
Title: A Phase 2 Clinical Trial Investigating the Effects of Obeticholic Acid on Lipoprotein Metabolism in Subjects With Primary Biliary Cirrhosis
Brief Title: Phase 2 Study on Effects of Obeticholic Acid (OCA) on Lipoprotein Metabolism in Participants With Primary Biliary Cirrhosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intercept Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 747-205
Record Dates: First submitted 2013-05-23; First posted 2013-05-31 (Estimated); Results first posted 2016-10-19 (Estimated); Last update posted 2022-08-24 (Actual); Status verified 2022-07

CONDITIONS: Primary Biliary Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — obeticholic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OCA: 10 mg (Experimental): Obeticholic acid, oral administration, 10 milligrams (mg), 8 weeks
  Interventions: Drug: Obeticholic Acid

INTERVENTIONS:
Drug: Obeticholic Acid — All participants were treated with OCA (oral administration, 10 mg, once daily [QD]) for 8 weeks and continued their prestudy dose of ursodeoxycholic acid (UDCA). After completion of the 8-week Primary Treatment Phase of the study and the 4-week follow-up period, during which time participants did not take OCA, all eligible participants were offered the opportunity to enter an open-label, long-term safety extension phase, during which they could receive 10 mg OCA QD for up to 2 years.
  Other Names: 6α-Ethyl chenodeoxycholic acid (6-ECDCA); INT-747

SUMMARY:
The purpose of this study was to determine if OCA had an effect on cholesterol levels in the blood in participants with primary biliary cirrhosis (PBC).

DETAILED DESCRIPTION:
This was a phase 2, open-label, multicenter study evaluating the effects of OCA on lipoprotein metabolism in participants with PBC; in particular, OCA's effects on high-density lipoprotein cholesterol. Nuclear magnetic resonance spectroscopy was utilized to quantify the changes in lipoprotein particle sizes and concentrations. Components of reverse cholesterol transport were also assessed.

ELIGIBILITY:
Key Inclusion Criteria:

1. Definite or probable PBC diagnosis as demonstrated by the presence of ≥ 2 of the following 3 diagnostic factors:

   * History of elevated alkaline phosphatase levels for at least 6 months
   * A positive anti-microbial antibody (AMA) titer or, if AMA negative or in low titer (<1:80), PBC-specific antibodies
   * Liver biopsy consistent with PBC
2. Taking UDCA for at least 12 months (stable dose for ≥ 3 months) prior to Day 0 or unable to tolerate UDCA (no UDCA for ≥ 3 months prior to Day 0).
3. Contraception: Female participants must have been postmenopausal, surgically sterile, or if premenopausal, were prepared to use ≥ 1 effective (≤ 1% failure rate) method of contraception during the trial and until at least 30 days after the last dose of Investigational Product.
4. Must have provided written informed consent and agreed to comply with the trial protocol.

Key Exclusion Criteria:

1. Participants with decompensated PBC (as determined by the Investigator).
2. Severe pruritus or systemic treatment for pruritus (for example, treatment with bile acid sequestrants or rifampicin) within 2 months of Day 0.
3. History or presence of other significant liver diseases including:

   * Active or chronic Hepatitis B or C virus infection
   * Primary sclerosing cholangitis
   * Alcoholic liver disease
   * Definite autoimmune liver disease or overlap hepatitis
   * Nonalcoholic steatohepatitis

   Note: Participants with Gilbert's disease or those with a history of hepatitis B who were currently antigen negative and seroconverted were not considered exclusionary.
4. Uncontrolled diabetes or other uncontrolled or unstable medical condition that may have interfered with trial results.
5. Administration of any of the following medications as specified below:

   * Prohibited 28 days prior to Day 0: bile acid sequestrants including cholestyramine, colesevelam, colestipol or omega-3 fatty acid containing dietary supplements
   * Prohibited 3 months prior to Day 0 and throughout trial participation: serum-lipid modifying agents including 3-hydroxy-3-methylglutaryl-coenzyme A reductase inhibitors, fenofibrate or other fibrates, nicotinic acid and derivatives, ezetimibe, Vitamin E (other than as standard dietary supplement)
   * Prohibited 6 months prior to Day 0 and throughout the trial participation: azathioprine, colchicine, cyclosporine, methotrexate, mycophenolate mofetil, pentoxifylline; budesonide and other systemic corticosteroids; potentially hepatotoxic drugs (including α-methyl-dopa, sodium valproic acid, isoniazide, or nitrofurantoin)
   * Prohibited 12 months prior to Day 0 and throughout the trial participation: antibodies or immunotherapy directed against interleukins or other cytokines or chemokines
6. Planned change in diet or exercise habits during participation in the trial.
7. Presence or history of clinically significant cardiac arrhythmias that may have prohibited the participant from participating in the trial.
8. If female: known pregnancy, or had a positive urine pregnancy test (confirmed by a positive serum pregnancy test), or lactating.
9. Recent (3 months prior to day 0) participation in another trial involving OCA or participation in another investigational trial (30 days prior to Day 0) and during the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-12-03 (Actual); Primary Completion 2014-08-13 (Actual); Study Completion 2016-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Harb, MD, Study Director — Intercept Pharmaceuticals, Inc.
Locations (7):
- United States (7):
  - Scripps Clinic, La Jolla, California
  - University of California, Davis Medical Center, Sacramento, California
  - University of Miami, Miami, Florida
  - Indiana University Medical Center, Indianapolis, Indiana
  - Beth Israel Medical Center, New York, New York
  - McGuire DVAMC, Richmond, Virginia
  - Swedish Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started 19-Nov-2013 and completed 16-May-2014 in the primary treatment phase (PTP). Thirty-three participants were screened and 27 enrolled.
Pre-assignment Details: Screening window was up to 20 days in duration to assess eligibility. Stable dose of ursodeoxycholic acid (UDCA) for 3 months prior to Day 0 was required. A 28-day washout period for bile acid sequestrants and no serum-lipid modifying agents for 3 months prior to Day 0 was also required. After the PTP, participants were offered the opportunity to enter the open-label, long-term safety extension (LTSE) phase of the study.
Groups:
- Primary Treatment Phase: All participants were treated with obeticholic acid (OCA) (oral administration, 10 milligrams [mg], once daily [QD]) for 8 weeks and continued their prestudy dose of UDCA. After completion of the 8-week PTP of the study and the 4-week follow-up period, during which time participants did not take OCA, all eligible participants were offered the opportunity to enter the open-label LTSE phase, during which they could receive 10 mg OCA QD for up to 2 years.
- Long-term Safety Extension Phase: Participants received OCA 10 mg QD for up to 2 years.
Period: Primary Treatment Phase
Arm/Group | Primary Treatment Phase | Long-term Safety Extension Phase
Started (One participant was thought to have been incorrectly dispensed 5-mg OCA during the PTP. This participant was not included in the ITT population and this participant's data was not included in any of the analyses.) | 27 | 0
Received at Least 1 Dose of Study Drug (One participant was thought to have been incorrectly dispensed 5-mg OCA during the PTP. This participant was not included in the ITT population and this participant's data was not included in any of the analyses.) | 27 | 0
Completed | 25 | 0
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0
Period: Long-term Safety Extension Phase
Arm/Group | Primary Treatment Phase | Long-term Safety Extension Phase
Started (Only eligible participants who completed the PTP phase enrolled in the LTSE phase.) | 0 (Only eligible participants who completed the PTP phase enrolled in the LTSE phase.) | 21 (Only eligible participants who completed the PTP phase enrolled in the LTSE phase.)
Received at Least 1 Dose of Study Drug | 0 | 21
Completed | 0 | 15
Not Completed | 0 | 6
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Pruritus | 0 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Participant Unavailable for Final Study Visit | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Obeticholic Acid: All participants were treated with OCA (oral administration, 10 mg, QD) for 8 weeks and continued their prestudy dose of UDCA. After completion of the 8-week PTP of the study and the 4-week follow-up period, during which time participants did not take OCA, eligible participants entered the open-label LTSE phase and received 10 mg OCA QD for up to 2 years.
Arm/Group | Obeticholic Acid
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (9.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 1
Race/Ethnicity, Customized [Number; unit: participants]
  White | 25
  Non-White/Hispanic | 1
Region of Enrollment [Number; unit: participants]
  United States | 26
High-density Lipoprotein (HDL) Cholesterol Concentration [Mean (Standard Deviation); unit: mmol/L] — Baseline measure reported in millimoles/liter (mmol/L).
  mmol/L | 1.86 (0.51798)
HDL Particle Size [Mean (Standard Deviation); unit: nm] — Baseline measure reported in nanometers (nm).
  nm | 10.19 (0.734)
HDL Particle Concentration (total) [Mean (Standard Deviation); unit: µmol/L] — Baseline measure reported in micromoles/L (umol/L).
  µmol/L | 30.08 (7.228)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline In High-density Lipoprotein (HDL) Cholesterol Concentration
Time Frame: Baseline, Week 8
Population: Intent-to-treat: all enrolled participants who received at least 1 dose of OCA during the study. All efficacy and safety endpoints were analyzed using the intent-to-treat population.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Groups:
- Primary Treatment Phase: All participants were treated with OCA (oral administration, 10 mg QD) for 8 weeks and continued their prestudy dose of UDCA. After completion of the 8-week PTP of the study and the 4-week follow-up period, during which time participants did not take OCA, all eligible participants were offered the opportunity to enter the open-label LTSE phase, during which they could receive 10 mg OCA QD for up to 2 years.
Arm/Group | Primary Treatment Phase
Number analyzed (Participants) | 23
mmol/L | -0.38 [-0.51 to -0.24]
Statistical Analysis 1: Comparison: Primary Treatment Phase; Test type: Superiority or Other; Mean Difference (Net) = -0.38, 95% CI 2-sided [-0.51 to -0.24]

2. Primary Outcome: Absolute Change From Baseline In HDL Particle Size
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: nm
Arm/Group | Primary Treatment Phase
Number analyzed (Participants) | 23
nm | -0.44 [-0.63 to -0.25]
Statistical Analysis 1: Comparison: Primary Treatment Phase; Test type: Superiority or Other; Mean Difference (Net) = -0.44, 95% CI 2-sided [-0.63 to -0.25]

3. Primary Outcome: Absolute Change From Baseline In HDL Particle Number
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: umol/L
Arm/Group | Primary Treatment Phase
Number analyzed (Participants) | 23
umol/L | -0.06 [-1.58 to 1.46]
Statistical Analysis 1: Comparison: Primary Treatment Phase; Test type: Superiority or Other; Mean Difference (Net) = -0.06, 95% CI 2-sided [-1.58 to 1.46]

4. Secondary Outcome: Median Change From Baseline In HDL Cholesterol Concentration At Weeks 4, 8, and 12
Time Frame: Baseline, Week 4, Week 8, Week 12
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Primary Treatment Phase
Number analyzed (Participants) | 26
mmol/L
  Week 4 | -0.2072 [-0.5957 to -0.0259]
  Week 8: number analyzed (Participants) | 23
  Week 8 | -0.3108 [-0.4403 to -0.0777]
  Week 12: number analyzed (Participants) | 25
  Week 12 | 0.0518 [-0.2849 to 0.1554]

5. Secondary Outcome: Median Change From Baseline In HDL Particle Size At Weeks 4, 8, and 12
Time Frame: Baseline, Week 4, Week 8, Week 12
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: nm
Arm/Group | Primary Treatment Phase
Number analyzed (Participants) | 26
nm
  Week 4 | -0.30 [-0.50 to -0.10]
  Week 8: number analyzed (Participants) | 23
  Week 8 | -0.30 [-0.60 to -0.10]
  Week 12: number analyzed (Participants) | 25
  Week 12 | 0.00 [-0.20 to 0.10]

6. Secondary Outcome: Median Change From Baseline In HDL Particle Number At Weeks 4, 8, and 12
Time Frame: Baseline, Week 4, Week 8, Week 12
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: umol/L
Arm/Group | Primary Treatment Phase
Number analyzed (Participants) | 26
umol/L
  Week 4 | 0.55 [-2.60 to 1.60]
  Week 8: number analyzed (Participants) | 23
  Week 8 | 0.60 [-1.60 to 1.70]
  Week 12: number analyzed (Participants) | 25
  Week 12 | 1.60 [-1.60 to 3.10]

7. Secondary Outcome: Median Change From Week 8 In HDL Cholesterol Concentration At Week 12
Time Frame: Week 8, Week 12
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Primary Treatment Phase
Number analyzed (Participants) | 22
mmol/L | 0.3108 [0.1036 to 0.5180]

8. Secondary Outcome: Median Change From Week 8 In HDL Particle Size At Week 12
Time Frame: Week 8, Week 12
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: nm
Arm/Group | Primary Treatment Phase
Number analyzed (Participants) | 22
nm | 0.30 [0.10 to 0.50]

9. Secondary Outcome: Median Change From Week 8 In HDL Particle Number At Week 12
Time Frame: Week 8, Week 12
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: umol/L
Arm/Group | Primary Treatment Phase
Number analyzed (Participants) | 22
umol/L | 1.40 [-0.60 to 3.10]

10. Secondary Outcome: Maximum Plasma Concentration (Cmax) Of OCA And Conjugates
Description: Results are reported in nanograms per milliliter (ng/mL).
Time Frame: Week 8
Population: The PK Population was comprised of all subjects who had at least 1 confirmed analyzable fasting sample at Week 8 and who did not have any major protocol deviations that potentially affected exposure levels. The PK Population was used for the OCA PK and bile acid analyses.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Primary Treatment Phase
Number analyzed (Participants) | 7
ng/mL
  OCA | 107 (112)
  Glycine Conjugate (Glyco)-OCA | 212 (144)
  Taurine Conjugate (Tauro)-OCA | 219 (208)
  Total-OCA | 409 (299)

11. Secondary Outcome: Time To Reach Cmax (Tmax) For OCA And Conjugates
Description: Results are reported in hours (h).
Time Frame: Week 8
Population: as for outcome 10
Measure: Median (Full Range); unit: h
Arm/Group | Primary Treatment Phase
Number analyzed (Participants) | 7
h
  OCA | 1.00 [0.750 to 4.00]
  Glyco-OCA | 5.00 [1.50 to 6.00]
  Tauro-OCA | 5.98 [5.00 to 6.00]
  Total-OCA | 5.00 [1.00 to 6.00]

12. Secondary Outcome: Area Under The Concentration-time Curve From Hour 0 To Last Sampling Time (Hour 6) (AUC0-6) For OCA And Conjugates
Description: Results are reported in hour*nanograms per milliliter (h*ng/mL).
Time Frame: Week 8
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Primary Treatment Phase
Number analyzed (Participants) | 7
h*ng/mL
  OCA | 189 (185)
  Glyco-OCA | 702 (644)
  Tauro-OCA | 698 (653)
  Total-OCA | 1360 (1150)

13. Secondary Outcome: Median Change From Baseline In Total Cholesterol
Time Frame: Baseline, Week 4, Week 8/End of Treatment (EOT), Week 12, Month 6, Month 12, Month 18, Month 24/EOT, Last Dose
Population: Intent-to-treat population, comprised of all enrolled participants who received at least 1 dose of OCA, was used for all efficacy and safety endpoints. The overall number of the participants is the total number of participants who had at least 1 lab measurement at any given timepoint, including the baseline. The number of participants at a given week may be smaller than the overall number of participants, because some patients may have no follow up measurement at that week, or no baseline.
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Primary Treatment Phase | Long-term Safety Extension Phase
Number analyzed (Participants) | 26 | 20
mmol/L
  Week 4: number analyzed (Participants) | 26 | 0
  Week 4 | -0.0518 [-0.8806 to 0.2590] |
  Week 8/EOT: number analyzed (Participants) | 23 | 0
  Week 8/EOT | -0.2849 [-0.7770 to 0.0777] |
  Week 12: number analyzed (Participants) | 25 | 0
  Week 12 | 0.2331 [-0.3885 to 0.4662] |
  Month 6: number analyzed (Participants) | 0 | 19
  Month 6 |  | -0.1813 [-0.8806 to 0.1295]
  Month 12: number analyzed (Participants) | 0 | 19
  Month 12 |  | 0.0777 [-0.1554 to 0.5698]
  Month 18: number analyzed (Participants) | 0 | 17
  Month 18 |  | 0.2849 [-0.2590 to 0.9842]
  Month 24/EOT: number analyzed (Participants) | 0 | 17
  Month 24/EOT |  | -0.0777 [-0.4144 to 0.2849]
  Last Dose: number analyzed (Participants) | 0 | 18
  Last Dose |  | 0.285 [-0.259 to 0.699]

14. Secondary Outcome: Median Change From Baseline In Total Triglycerides
Time Frame: Baseline, Week 4, Week 8/End of Treatment (EOT), Week 12, Month 6, Month 12, Month 18, Month 24/EOT, Last Dose
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Primary Treatment Phase | Long-term Safety Extension Phase
Number analyzed (Participants) | 26 | 20
mmol/L
  Week 4: number analyzed (Participants) | 26 | 0
  Week 4 | -0.0226 [-0.2260 to 0.0678] |
  Week 8/EOT: number analyzed (Participants) | 23 | 0
  Week 8/EOT | 0.0565 [-0.1130 to 0.2373] |
  Week 12: number analyzed (Participants) | 25 | 0
  Week 12 | 0.1130 [-0.0113 to 0.2147] |
  Month 6: number analyzed (Participants) | 0 | 19
  Month 6 |  | -0.1469 [-0.4633 to 0.0791]
  Month 12: number analyzed (Participants) | 0 | 19
  Month 12 |  | -0.0113 [-0.2938 to 0.2260]
  Month 18: number analyzed (Participants) | 0 | 17
  Month 18 |  | -0.0565 [-0.2034 to 0.2260]
  Month 24/EOT: number analyzed (Participants) | 0 | 17
  Month 24/EOT |  | 0.000 [-0.2260 to 0.1130]
  Last Dose: number analyzed (Participants) | 0 | 18
  Last Dose |  | -0.068 [-0.260 to 0.226]

15. Secondary Outcome: Median Change From Baseline In Low-density Lipoprotein (LDL) Cholesterol (Direct)
Time Frame: Baseline, Week 4, Week 8/End of Treatment (EOT), Week 12, Month 6, Month 12, Month 18, Month 24/EOT, Last Dose
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Primary Treatment Phase | Long-term Safety Extension Phase
Number analyzed (Participants) | 26 | 20
mmol/L
  Week 4: number analyzed (Participants) | 26 | 0
  Week 4 | 0.27 [0.21 to 0.36] |
  Week 8/EOT: number analyzed (Participants) | 23 | 0
  Week 8/EOT | 0.31 [0.05 to 0.41] |
  Week 12: number analyzed (Participants) | 25 | 0
  Week 12 | 0.18 [-0.21 to 0.39] |
  Month 6: number analyzed (Participants) | 0 | 19
  Month 6 |  | 0.3108 [-0.0777 to 0.6216]
  Month 12: number analyzed (Participants) | 0 | 19
  Month 12 |  | 0.4403 [0.1036 to 0.7511]
  Month 18: number analyzed (Participants) | 0 | 17
  Month 18 |  | 0.5957 [0.1813 to 1.0360]
  Month 24/EOT: number analyzed (Participants) | 0 | 17
  Month 24/EOT |  | 0.3108 [0.1295 to 0.6216]
  Last Dose: number analyzed (Participants) | 0 | 18
  Last Dose |  | 0.518 [0.233 to 0.648]

16. Secondary Outcome: Median Change From Baseline In LDL Particle Size
Time Frame: Baseline, Week 4, Week 8/End of Treatment (EOT), Week 12, Month 6, Month 12, Month 18, Month 24/EOT, Last Dose
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: nm
Arm/Group | Primary Treatment Phase | Long-term Safety Extension Phase
Number analyzed (Participants) | 26 | 20
nm
  Week 4: number analyzed (Participants) | 26 | 0
  Week 4 | -0.30 [-0.50 to -0.10] |
  Week 8/EOT: number analyzed (Participants) | 23 | 0
  Week 8/EOT | -0.10 [-0.40 to 0.10] |
  Week 12: number analyzed (Participants) | 25 | 0
  Week 12 | 0.00 [-0.30 to 0.20] |
  Month 6: number analyzed (Participants) | 0 | 19
  Month 6 |  | -0.10 [-0.30 to 0.30]
  Month 12: number analyzed (Participants) | 0 | 19
  Month 12 |  | -0.20 [-0.50 to 0.30]
  Month 18: number analyzed (Participants) | 0 | 17
  Month 18 |  | -0.10 [-0.50 to 0.10]
  Month 24/EOT: number analyzed (Participants) | 0 | 17
  Month 24/EOT |  | -0.10 [-0.20 to 0.20]
  Last Dose: number analyzed (Participants) | 0 | 18
  Last Dose |  | -0.10 [-0.50 to 0.10]

17. Secondary Outcome: Median Change From Baseline In Total LDL Particles
Description: Results are reported in nanomoles per liter (nmol/L).
Time Frame: Baseline, Week 4, Week 8/End of Treatment (EOT), Week 12, Month 6, Month 12, Month 18, Month 24/EOT, Last Dose
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | Primary Treatment Phase | Long-term Safety Extension Phase
Number analyzed (Participants) | 26 | 20
nmol/L
  Week 4: number analyzed (Participants) | 26 | 0
  Week 4 | 108.0 [73.0 to 231.0] |
  Week 8/EOT: number analyzed (Participants) | 23 | 0
  Week 8/EOT | 128.0 [57.0 to 273.0] |
  Week 12: number analyzed (Participants) | 25 | 0
  Week 12 | 159.0 [18.0 to 197.0] |
  Month 6 (Small): number analyzed (Participants) | 0 | 19
  Month 6 (Small) |  | 148.0 [-17.0 to 295.0]
  Month 12 (Small): number analyzed (Participants) | 0 | 19
  Month 12 (Small) |  | 89.0 [-13.0 to 318.0]
  Month 18 (Small): number analyzed (Participants) | 0 | 17
  Month 18 (Small) |  | 18.0 [-15.0 to 261.0]
  Month 24/EOT (Small): number analyzed (Participants) | 0 | 17
  Month 24/EOT (Small) |  | 34.0 [-5.0 to 74.0]
  Last Dose (Small): number analyzed (Participants) | 0 | 18
  Last Dose (Small) |  | 22.0 [-23.0 to 98.0]
  Month 6 (Large): number analyzed (Participants) | 0 | 19
  Month 6 (Large) |  | 9.0 [-102.0 to 138.0]
  Month 12 (Large): number analyzed (Participants) | 0 | 19
  Month 12 (Large) |  | -53.0 [-190.0 to 155.0]
  Month 18 (Large): number analyzed (Participants) | 0 | 17
  Month 18 (Large) |  | -18.0 [-199.0 to 143.0]
  Month 24/EOT (Large): number analyzed (Participants) | 0 | 17
  Month 24/EOT (Large) |  | -122.0 [-229.0 to 60.0]
  Last Dose (Large): number analyzed (Participants) | 0 | 18
  Last Dose (Large) |  | -8.0 [-243.0 to 162.0]
  Month 6 (Intermediate-density Lipoprotein [IDL]): number analyzed (Participants) | 0 | 19
  Month 6 (Intermediate-density Lipoprotein [IDL]) |  | -12.0 [-121.0 to 72.0]
  Month 12 (IDL): number analyzed (Participants) | 0 | 19
  Month 12 (IDL) |  | -57.0 [-117.0 to 21.0]
  Month 18 (IDL): number analyzed (Participants) | 0 | 17
  Month 18 (IDL) |  | -43.0 [-104.0 to 112.0]
  Month 24/EOT (IDL): number analyzed (Participants) | 0 | 17
  Month 24/EOT (IDL) |  | 78.0 [-17.0 to 151.0]
  Last Dose (IDL): number analyzed (Participants) | 0 | 18
  Last Dose (IDL) |  | 11.0 [-89.0 to 129.0]

18. Secondary Outcome: Median Change From Baseline In Very Low-density Lipoprotein (VLDL) Cholesterol
Description: Results are reported in milligrams per deciliter (mg/dL).
Time Frame: Baseline, Week 12, Month 6, Month 12, Month 18, Month 24/EOT, Last Dose
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: mg/dL
Arm/Group | Primary Treatment Phase | Long-term Safety Extension Phase
Number analyzed (Participants) | 25 | 20
mg/dL
  Week 12: number analyzed (Participants) | 25 | 0
  Week 12 | 5.0 [-3.0 to 7.0] |
  Month 6: number analyzed (Participants) | 0 | 19
  Month 6 |  | -21.0 [-41.0 to 7.0]
  Month 12: number analyzed (Participants) | 0 | 19
  Month 12 |  | -7.0 [-29.0 to 7.0]
  Month 18: number analyzed (Participants) | 0 | 17
  Month 18 |  | -14.0 [-25.0 to 3.0]
  Month 24/EOT: number analyzed (Participants) | 0 | 17
  Month 24/EOT |  | -1.0 [-8.0 to 15.0]
  Last Dose: number analyzed (Participants) | 0 | 18
  Last Dose |  | -11.5 [-29.0 to 3.0]

19. Secondary Outcome: Median Change From Baseline In VLDL Particle Size
Time Frame: Baseline, Week 4, Week 8/End of Treatment (EOT), Week 12, Month 6, Month 12, Month 18, Month 24/EOT, Last Dose
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: nm
Arm/Group | Primary Treatment Phase | Long-term Safety Extension Phase
Number analyzed (Participants) | 26 | 21
nm
  Week 4: number analyzed (Participants) | 24 | 0
  Week 4 | 42.55 [39.20 to 44.75] |
  Week 8/EOT: number analyzed (Participants) | 19 | 0
  Week 8/EOT | 43.40 [39.70 to 45.90] |
  Week 12: number analyzed (Participants) | 23 | 0
  Week 12 | 45.10 [43.30 to 48.40] |
  Month 6: number analyzed (Participants) | 0 | 15
  Month 6 |  | -4.80 [-9.50 to 0.90]
  Month 12: number analyzed (Participants) | 0 | 17
  Month 12 |  | -3.50 [-8.20 to 0.50]
  Month 18: number analyzed (Participants) | 0 | 15
  Month 18 |  | -4.90 [-6.00 to 2.90]
  Month 24/EOT: number analyzed (Participants) | 0 | 16
  Month 24/EOT |  | 0.50 [-2.05 to 5.20]
  Last Dose: number analyzed (Participants) | 0 | 16
  Last Dose |  | -4.10 [-5.95 to 1.75]

20. Secondary Outcome: Median Change From Baseline In VLDL Particles
Time Frame: Baseline, Week 4, Week 8/End of Treatment (EOT), Week 12, Month 6, Month 12, Month 18, Month 24/EOT, Last Dose
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | Primary Treatment Phase | Long-term Safety Extension Phase
Number analyzed (Participants) | 26 | 21
nmol/L
  Week 4: number analyzed (Participants) | 26 | 0
  Week 4 | -5.55 [-17.20 to -1.60] |
  Week 8/EOT: number analyzed (Participants) | 23 | 0
  Week 8/EOT | 2.70 [-14.80 to 9.10] |
  Week 12: number analyzed (Participants) | 25 | 0
  Week 12 | -0.90 [-9.50 to 10.90] |
  Month 6: number analyzed (Participants) | 0 | 19
  Month 6 |  | -4.70 [-34.50 to 9.50]
  Month 12: number analyzed (Participants) | 0 | 19
  Month 12 |  | -6.20 [-27.90 to 19.20]
  Month 18: number analyzed (Participants) | 0 | 17
  Month 18 |  | -6.80 [-25.10 to 0.30]
  Month 24/EOT: number analyzed (Participants) | 0 | 17
  Month 24/EOT |  | -0.30 [-16.10 to 12.60]
  Last Dose: number analyzed (Participants) | 0 | 18
  Last Dose |  | -6.80 [-19.00 to 6.20]

21. Secondary Outcome: Median Change From Baseline In Apolipoprotein A1 (ApoA1)
Description: Results are reported in grams per liter (g/L).
Time Frame: Baseline, Week 4, Week 8/End of Treatment (EOT), Week 12, Month 6, Month 12, Month 18, Month 24/EOT, Last Dose
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: g/L
Arm/Group | Primary Treatment Phase | Long-term Safety Extension Phase
Number analyzed (Participants) | 26 | 21
g/L
  Week 4: number analyzed (Participants) | 26 | 00
  Week 4 | -0.1000 [-0.1600 to 0.0000] |
  Week 8/EOT: number analyzed (Participants) | 23 | 0
  Week 8/EOT | -0.0600 [-0.2700 to 0.0000] |
  Week 12: number analyzed (Participants) | 25 | 0
  Week 12 | 0.0400 [-0.0200 to 0.1500] |
  Month 6: number analyzed (Participants) | 0 | 19
  Month 6 |  | -0.1400 [-0.2100 to 0.0700]
  Month 12: number analyzed (Participants) | 0 | 19
  Month 12 |  | -0.0900 [-0.2000 to 0.0100]
  Month 18: number analyzed (Participants) | 0 | 17
  Month 18 |  | -0.1000 [-0.1800 to 0.0300]
  Month 24/EOT: number analyzed (Participants) | 0 | 17
  Month 24/EOT |  | 0.0100 [-0.0600 to 0.0700]
  Last Dose: number analyzed (Participants) | 0 | 18
  Last Dose |  | -0.045 [-0.170 to 0.030]

22. Secondary Outcome: Median Change From Baseline In Apolipoprotein B (ApoB)
Time Frame: Baseline, Week 4, Week 8/End of Treatment (EOT), Week 12, Month 6, Month 12, Month 18, Month 24/EOT, Last Dose
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Primary Treatment Phase | Long-term Safety Extension Phase
Number analyzed (Participants) | 26 | 20
units on a scale
  Week 4: number analyzed (Participants) | 26 | 0
  Week 4 | 0.0950 [-0.0300 to 0.1200] |
  Week 8/EOT: number analyzed (Participants) | 23 | 0
  Week 8/EOT | 0.0700 [0.0000 to 0.1200] |
  Week 12: number analyzed (Participants) | 25 | 0
  Week 12 | 0.0500 [-0.0400 to 0.1000] |
  Month 6: number analyzed (Participants) | 0 | 19
  Month 6 |  | 0.0400 [0.0100 to 0.1100]
  Month 12: number analyzed (Participants) | 0 | 19
  Month 12 |  | 0.0400 [-0.0200 to 0.1000]
  Month 18: number analyzed (Participants) | 0 | 17
  Month 18 |  | 0.0600 [0.0400 to 0.1700]
  Month 24/EOT: number analyzed (Participants) | 0 | 17
  Month 24/EOT |  | 0.0900 [0.0300 to 0.1500]
  Last Dose: number analyzed (Participants) | 0 | 18
  Last Dose |  | 0.060 [0.040 to 0.170]

23. Secondary Outcome: Median Change From Baseline In ApoA1/ApoB Ratio
Time Frame: Baseline, Week 12, Month 6, Month 12, Month 18, Month 24/EOT, Last Dose
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Primary Treatment Phase | Long-term Safety Extension Phase
Number analyzed (Participants) | 25 | 20
Ratio
  Week 12: number analyzed (Participants) | 25 | 0
  Week 12 | -0.0503 [-0.1856 to 0.1939] |
  Month 6: number analyzed (Participants) | 0 | 19
  Month 6 |  | -0.2174 [-0.3638 to -0.0775]
  Month 12: number analyzed (Participants) | 0 | 19
  Month 12 |  | -0.1659 [-0.4509 to -0.0352]
  Month 18: number analyzed (Participants) | 0 | 17
  Month 18 |  | -0.2860 [-0.3918 to -0.0206]
  Month 24/EOT: number analyzed (Participants) | 0 | 17
  Month 24/EOT |  | -0.1172 [-0.3060 to 0.1613]
  Last Dose: number analyzed (Participants) | 0 | 18
  Last Dose |  | -0.291 [-0.390 to 0.015]

24. Secondary Outcome: Median Change From Baseline In Apolipoprotein E
Time Frame: Baseline, Week 4, Week 8/End of Treatment (EOT), Week 12, Month 6, Month 12, Month 18, Month 24/EOT, Last Dose
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Primary Treatment Phase | Long-term Safety Extension Phase
Number analyzed (Participants) | 25 | 20
mg/dL
  Week 4: number analyzed (Participants) | 24 | 0
  Week 4 | -0.85 [-1.80 to 0.20] |
  Week 8/EOT: number analyzed (Participants) | 22 | 0
  Week 8/EOT | -0.65 [-2.10 to 0.30] |
  Week 12: number analyzed (Participants) | 14 | 0
  Week 12 | 0.50 [-1.00 to 1.20] |
  Month 6: number analyzed (Participants) | 0 | 19
  Month 6 |  | -0.30 [-1.00 to 0.30]
  Month 12: number analyzed (Participants) | 0 | 19
  Month 12 |  | -0.30 [-0.80 to 0.50]
  Month 18: number analyzed (Participants) | 0 | 17
  Month 18 |  | -0.10 [-0.70 to 0.30]
  Month 24/EOT: number analyzed (Participants) | 0 | 17
  Month 24/EOT |  | 0.00 [-0.60 to 1.00]
  Last Dose: number analyzed (Participants) | 0 | 18
  Last Dose |  | 0.00 [-0.70 to 0.50]

25. Secondary Outcome: Median Change From Baseline In Lipoprotein-a
Time Frame: Baseline, Week 4, Week 8/End of Treatment (EOT), Week 12, Month 6, Month 12, Month 18, Month 24/EOT, Last Dose
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: umol/L
Arm/Group | Primary Treatment Phase | Long-term Safety Extension Phase
Number analyzed (Participants) | 26 | 20
umol/L
  Week 4: number analyzed (Participants) | 26 | 0
  Week 4 | 0.0000 [-0.0714 to 0.0000] |
  Week 8/EOT: number analyzed (Participants) | 23 | 0
  Week 8/EOT | 0.0000 [-0.0571 to 0.0000] |
  Week 12: number analyzed (Participants) | 25 | 0
  Week 12 | 0.0000 [-0.0357 to 0.0357] |
  Month 6: number analyzed (Participants) | 0 | 19
  Month 6 |  | 0.0000 [-0.0571 to 0.0357]
  Month 12: number analyzed (Participants) | 0 | 19
  Month 12 |  | 0.0000 [-0.0357 to 0.0357]
  Month 18: number analyzed (Participants) | 0 | 17
  Month 18 |  | 0.0000 [-0.0357 to 0.0000]
  Month 24/EOT: number analyzed (Participants) | 0 | 17
  Month 24/EOT |  | 0.0000 [-0.0286 to 0.0107]
  Last Dose: number analyzed (Participants) | 0 | 18
  Last Dose |  | 0.000 [-0.036 to 0.000]

26. Secondary Outcome: Median Change From Baseline In Lecithin-cholesterol Acyltransferase Activity
Description: Results are reported in nanomoles/milliliter/hour (nmol/mL/h).
Time Frame: Baseline, Week 4, Week 8/End of Treatment (EOT), Week 12, Month 6, Month 12, Month 18, Month 24/EOT
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: nmol/mL/h
Arm/Group | Primary Treatment Phase | Long-term Safety Extension Phase
Number analyzed (Participants) | 26 | 20
nmol/mL/h
  Week 4: number analyzed (Participants) | 24 | 0
  Week 4 | -20.5 [-74.5 to 21.5] |
  Week 8/EOT: number analyzed (Participants) | 22 | 0
  Week 8/EOT | -13.5 [-87.5 to 18.0] |
  Week 12: number analyzed (Participants) | 14 | 0
  Week 12 | 15.5 [-1.0 to 61.0] |
  Month 6: number analyzed (Participants) | 0 | 19
  Month 6 |  | -47.0 [-107.0 to 49.0]
  Month 12: number analyzed (Participants) | 0 | 19
  Month 12 |  | 46.0 [-29.0 to 75.0]
  Month 18: number analyzed (Participants) | 0 | 17
  Month 18 |  | -19.0 [-87.0 to 55.0]
  Month 24/EOT: number analyzed (Participants) | 0 | 17
  Month 24/EOT |  | -56.0 [-105.0 to -28.0]

27. Secondary Outcome: Median Change From Baseline In Cholesteryl Ester Transfer Protein
Description: Results are reported in picomole/milliliter/minute (pmol/mL/min).
Time Frame: Baseline, Week 4, Week 8/End of Treatment (EOT), Week 12, Month 6, Month 12, Month 18, Month 24/EOT
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: pmol/mL/min
Arm/Group | Primary Treatment Phase | Long-term Safety Extension Phase
Number analyzed (Participants) | 26 | 20
pmol/mL/min
  Week 4: number analyzed (Participants) | 24 | 0
  Week 4 | 1.95 [-0.25 to 3.25] |
  Week 8/EOT: number analyzed (Participants) | 22 | 0
  Week 8/EOT | 0.30 [-2.70 to 3.20] |
  Week 12: number analyzed (Participants) | 14 | 0
  Week 12 | 4.70 [1.80 to 10.10] |
  Month 6: number analyzed (Participants) | 0 | 19
  Month 6 |  | 1.20 [-1.40 to 4.40]
  Month 12: number analyzed (Participants) | 0 | 19
  Month 12 |  | -0.60 [-2.70 to 2.50]
  Month 18: number analyzed (Participants) | 0 | 17
  Month 18 |  | 0.50 [-1.00 to 4.50]
  Month 24/EOT: number analyzed (Participants) | 0 | 17
  Month 24/EOT |  | 0.40 [-3.70 to 4.70]

28. Secondary Outcome: Median Change From Baseline In Prebeta-1 HDL Concentration
Description: Results are reported in microgram/milliliter (ug/mL).
Time Frame: Baseline, Week 4, Week 8/End of Treatment (EOT), Month 6, Month 12, Month 18, Month 24/EOT
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: ug/mL
Arm/Group | Primary Treatment Phase | Long-term Safety Extension Phase
Number analyzed (Participants) | 26 | 18
ug/mL
  Week 4: number analyzed (Participants) | 24 | 0
  Week 4 | 1.55 [-11.50 to 11.45] |
  Week 8: number analyzed (Participants) | 20 | 0
  Week 8 | 7.55 [-7.35 to 58.85] |
  Month 6: number analyzed (Participants) | 0 | 15
  Month 6 |  | -6.90 [-22.00 to 9.00]
  Month 12: number analyzed (Participants) | 0 | 16
  Month 12 |  | -10.05 [-31.95 to 5.37]
  Month 18: number analyzed (Participants) | 0 | 9
  Month 18 |  | 1.94 [-6.80 to 4.30]
  Month 24/EOT: number analyzed (Participants) | 0 | 12
  Month 24/EOT |  | -1.35 [-5.90 to 3.07]

29. Secondary Outcome: Median Change From Baseline In Macrophage Cholesterol Efflux
Description: Results are reported as a percentage of cholesterol.
Time Frame: Baseline, Week 4, Week 8/End of Treatment (EOT), Month 6, Month 12, Month 18, Month 24/EOT
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: percentage of cholesterol
Arm/Group | Primary Treatment Phase | Long-term Safety Extension Phase
Number analyzed (Participants) | 25 | 20
percentage of cholesterol
  Week 4: number analyzed (Participants) | 24 | 0
  Week 4 | -0.800 [-2.465 to 0.120] |
  Week 8: number analyzed (Participants) | 22 | 0
  Week 8 | -0.705 [-1.240 to 0.350] |
  Month 6: number analyzed (Participants) | 0 | 16
  Month 6 |  | -1.745 [-3.170 to -0.140]
  Month 12: number analyzed (Participants) | 0 | 16
  Month 12 |  | -1.940 [-3.110 to 0.160]
  Month 18: number analyzed (Participants) | 0 | 13
  Month 18 |  | -2.450 [-3.500 to -0.680]
  Month 24/EOT: number analyzed (Participants) | 0 | 14
  Month 24/EOT |  | -0.770 [-2.610 to 0.580]

30. Secondary Outcome: Median Change From Baseline In C-reactive Protein
Time Frame: Baseline, Week 4, Week 8/End of Treatment (EOT), Week 12, Month 6, Month 12, Month 18, Month 24/EOT
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | Primary Treatment Phase | Long-term Safety Extension Phase
Number analyzed (Participants) | 23 | 20
nmol/L
  Week 4: number analyzed (Participants) | 14 | 0
  Week 4 | 0.0000 [0.0000 to 12.3812] |
  Week 8/EOT: number analyzed (Participants) | 15 | 0
  Week 8/EOT | 0.0000 [-9.5340 to 4.7620] |
  Week 12: number analyzed (Participants) | 15 | 0
  Week 12 | 11.4288 [0.0000 to 28.5720] |
  Month 6: number analyzed (Participants) | 0 | 19
  Month 6 |  | 0.00 [-4.76 to 0.00]
  Month 12: number analyzed (Participants) | 0 | 19
  Month 12 |  | 0.00 [-4.76 to 0.00]
  Month 18: number analyzed (Participants) | 0 | 17
  Month 18 |  | 0.00 [-4.76 to 0.00]
  Month 24/EOT: number analyzed (Participants) | 0 | 16
  Month 24/EOT |  | 0.00 [0.00 to 0.00]

31. Secondary Outcome: Median Change From Baseline In Glycoprotein A
Description: Results are reported in picograms/milliliter (pg/mL).
Time Frame: Baseline, Week 12, Month 6, Month 12, Month 18, Month 24/EOT
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Primary Treatment Phase | Long-term Safety Extension Phase
Number analyzed (Participants) | 25 | 20
pg/mL
  Week 12: number analyzed (Participants) | 25 | 0
  Week 12 | 12.0 [-6.0 to 36.0] |
  Month 6: number analyzed (Participants) | 0 | 19
  Month 6 |  | -27.0 [-54.0 to 15.0]
  Month 12: number analyzed (Participants) | 0 | 19
  Month 12 |  | -13.0 [-61.0 to 10.0]
  Month 18: number analyzed (Participants) | 0 | 17
  Month 18 |  | -26.0 [-41.0 to 19.0]
  Month 24/EOT: number analyzed (Participants) | 0 | 17
  Month 24/EOT |  | 10.0 [-10.0 to 48.0]

32. Secondary Outcome: Median Change From Baseline In Fibroblast Growth Factor-19
Time Frame: Baseline, Week 4, Week 8/End of Treatment (EOT), Week 12, Month 6, Month 12, Month 18, Month 24/EOT
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Primary Treatment Phase | Long-term Safety Extension Phase
Number analyzed (Participants) | 25 | 20
pg/mL
  Week 4: number analyzed (Participants) | 25 | 0
  Week 4 | 81.8800 [-25.5290 to 316.0650] |
  Week 8/EOT: number analyzed (Participants) | 23 | 0
  Week 8/EOT | 112.5460 [36.5310 to 226.1710] |
  Week 12: number analyzed (Participants) | 24 | 0
  Week 12 | 16.8400 [-35.4980 to 30.6920] |
  Month 6: number analyzed (Participants) | 0 | 19
  Month 6 |  | 81.390 [-6.600 to 201.000]
  Month 12: number analyzed (Participants) | 0 | 19
  Month 12 |  | 29.220 [-49.190 to 144.350]
  Month 18: number analyzed (Participants) | 0 | 17
  Month 18 |  | 55.230 [4.320 to 127.290]
  Month 24/EOT: number analyzed (Participants) | 0 | 17
  Month 24/EOT |  | -0.740 [-53.770 to 22.910]

33. Secondary Outcome: Participants With Lipoprotein X
Description: Lipoprotein samples were assessed using nuclear magnetic resonance spectroscopy for the presence/absence of Lipoprotein X. Lipoprotein X sometimes appears with advanced cholestasis and can confound assessment of other lipoprotein concentrations, particularly LDL.
Time Frame: Week 12 and Last Dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Treatment Phase | Long-term Safety Extension Phase
Number analyzed (Participants) | 26 | 21
Participants
  Week 12 | 1 | 0
  Last Dose | 0 | 0

34. Secondary Outcome: Median Change From Baseline In Alkaline Phosphatase
Description: Results are reported in units/Liter (U/L).
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24/EOT
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Long-term Safety Extension Phase
Number analyzed (Participants) | 20
U/L
  Month 6: number analyzed (Participants) | 19
  Month 6 | -43.40 [-87.10 to -13.10]
  Month 12: number analyzed (Participants) | 19
  Month 12 | -31.50 [-69.90 to -6.70]
  Month 18: number analyzed (Participants) | 17
  Month 18 | -31.90 [-47.20 to 1.70]
  Month 24/EOT: number analyzed (Participants) | 16
  Month 24/EOT | 6.40 [-28.75 to 38.05]

35. Secondary Outcome: Median Change From Baseline In Gamma-glutamyl Transferase
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24/EOT
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Long-term Safety Extension Phase
Number analyzed (Participants) | 20
U/L
  Month 6: number analyzed (Participants) | 19
  Month 6 | -59.40 [-80.90 to -21.30]
  Month 12: number analyzed (Participants) | 19
  Month 12 | -41.60 [-92.30 to -28.30]
  Month 18: number analyzed (Participants) | 17
  Month 18 | -40.80 [-90.80 to -27.70]
  Month 24/EOT: number analyzed (Participants) | 16
  Month 24/EOT | -30.05 [-49.50 to 6.35]

36. Secondary Outcome: Median Change From Baseline In Alanine Aminotransferase
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24/EOT
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Long-term Safety Extension Phase
Number analyzed (Participants) | 20
U/L
  Month 6: number analyzed (Participants) | 19
  Month 6 | -9.80 [-15.90 to -3.60]
  Month 12: number analyzed (Participants) | 19
  Month 12 | -9.80 [-16.20 to -1.00]
  Month 18: number analyzed (Participants) | 17
  Month 18 | -11.80 [-25.00 to -3.40]
  Month 24/EOT: number analyzed (Participants) | 16
  Month 24/EOT | -5.95 [-14.85 to 7.95]

37. Secondary Outcome: Median Change From Baseline In Aspartate Aminotransferase
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24/EOT
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Long-term Safety Extension Phase
Number analyzed (Participants) | 20
U/L
  Month 6: number analyzed (Participants) | 19
  Month 6 | -5.30 [-15.00 to -1.40]
  Month 12: number analyzed (Participants) | 19
  Month 12 | -3.60 [-8.20 to 1.60]
  Month 18: number analyzed (Participants) | 17
  Month 18 | -6.00 [-18.60 to -1.70]
  Month 24/EOT: number analyzed (Participants) | 16
  Month 24/EOT | -4.50 [-13.50 to 4.00]

38. Secondary Outcome: Median Change From Baseline In Total And Unconjugated (Direct) Bilirubin
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24/EOT
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: umol/L
Arm/Group | Long-term Safety Extension Phase
Number analyzed (Participants) | 20
umol/L
  Month 6: number analyzed (Participants) | 19
  Month 6 | 0.0000 [0.0000 to 0.0000]
  Month 12: number analyzed (Participants) | 19
  Month 12 | 0.0000 [0.0000 to 0.0000]
  Month 18: number analyzed (Participants) | 17
  Month 18 | 0.0000 [0.0000 to 0.0000]
  Month 24/EOT: number analyzed (Participants) | 16
  Month 24/EOT | 0.0000 [0.0000 to 0.0000]

39. Secondary Outcome: Median Change From Baseline In Albumin
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24/EOT
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: g/L
Arm/Group | Long-term Safety Extension Phase
Number analyzed (Participants) | 20
g/L
  Month 6: number analyzed (Participants) | 19
  Month 6 | -0.60 [-1.80 to 3.20]
  Month 12: number analyzed (Participants) | 19
  Month 12 | -0.20 [-2.10 to 3.20]
  Month 18: number analyzed (Participants) | 17
  Month 18 | 1.30 [0.30 to 4.30]
  Month 24/EOT: number analyzed (Participants) | 16
  Month 24/EOT | 0.05 [-1.40 to 3.75]

40. Secondary Outcome: Median Change From Baseline In Prothrombin Time
Description: Results are reported in seconds (sec).
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24/EOT
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: sec
Arm/Group | Long-term Safety Extension Phase
Number analyzed (Participants) | 20
sec
  Month 6: number analyzed (Participants) | 19
  Month 6 | 0.000 [-0.500 to 0.900]
  Month 12: number analyzed (Participants) | 18
  Month 12 | -0.050 [-0.600 to 0.400]
  Month 18: number analyzed (Participants) | 17
  Month 18 | 0.400 [0.100 to 0.800]
  Month 24/EOT: number analyzed (Participants) | 16
  Month 24/EOT | 0.200 [-0.200 to 0.750]

41. Secondary Outcome: Median Change From Baseline In Prothrombin International Normalized Ratio
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24/EOT
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Long-term Safety Extension Phase
Number analyzed (Participants) | 20
ratio
  Month 6: number analyzed (Participants) | 19
  Month 6 | 0.0000 [0.0000 to 0.1000]
  Month 12: number analyzed (Participants) | 18
  Month 12 | 0.0000 [0.0000 to 0.0000]
  Month 18: number analyzed (Participants) | 17
  Month 18 | 0.0000 [0.0000 to 0.1000]
  Month 24/EOT: number analyzed (Participants) | 16
  Month 24/EOT | 0.0000 [0.0000 to 0.0500]

42. Secondary Outcome: Median Change From Baseline In Enhanced Liver Fibrosis (ELF) Score
Description: Change in ELF was calculated as ELF score at the end of the study minus ELF score prior to the intervention (at baseline). A decrease in the ELF score was considered good as it reflected a decrease in liver fibrosis, and an increase in ELF score was considered bad as it reflected an increase in liver fibrosis.
  Change in ELF scores ranged from -0.56 (good) to + 0.68 (bad).
Time Frame: Baseline, Month 12, Month 24/EOT
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Long-term Safety Extension Phase
Number analyzed (Participants) | 20
score on a scale
  Month 12: number analyzed (Participants) | 19
  Month 12 | 0.000 [-0.300 to 0.500]
  Week 24/EOT: number analyzed (Participants) | 16
  Week 24/EOT | 0.150 [-0.050 to 0.550]

43. Secondary Outcome: Median Change From Baseline In Hyaluronic Acid
Time Frame: Baseline, Month 12, Month 24/EOT
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Long-term Safety Extension Phase
Number analyzed (Participants) | 20
ng/mL
  Month 12: number analyzed (Participants) | 19
  Month 12 | -5.700 [-21.020 to 15.770]
  Month 24/EOT: number analyzed (Participants) | 16
  Month 24/EOT | -1.805 [-16.665 to 17.830]

44. Secondary Outcome: Median Change From Baseline In Amino-terminal Propeptide Of Type III Procollagen
Description: Results are reported in micrograms/Liter (ug/L).
Time Frame: Baseline, Month 12, Month 24/EOT
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ug/L
Arm/Group | Long-term Safety Extension Phase
Number analyzed (Participants) | 20
ug/L
  Month 12: number analyzed (Participants) | 19
  Month 12 | 0.670 [-0.220 to 1.200]
  Month 24/EOT: number analyzed (Participants) | 16
  Month 24/EOT | 2.095 [1.010 to 3.310]

45. Secondary Outcome: Median Change From Baseline In Tissue Inhibitor Of Metalloproteinases 1
Time Frame: Baseline, Month 12, Month 24/EOT
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ug/L
Arm/Group | Long-term Safety Extension Phase
Number analyzed (Participants) | 20
ug/L
  Month 12: number analyzed (Participants) | 19
  Month 12 | 9.600 [-15.700 to 16.600]
  Month 24/EOT: number analyzed (Participants) | 16
  Month 24/EOT | 2.000 [-14.300 to 23.650]

46. Secondary Outcome: Median Change From Baseline In Hepatic Stiffness
Description: Results are reported in kilopascal (kPa).
Time Frame: Baseline, Month 12, Month 24/EOT
Population: Intent-to-treat was comprised of all enrolled participants who received at least 1 dose of OCA during the study. All efficacy and safety endpoints were analyzed using the intent-to-treat population. The number of participants analyzed includes the subjects who were available at the specific time point of analysis.
Measure: Median (Inter-Quartile Range); unit: kPa
Arm/Group | Long-term Safety Extension Phase
Number analyzed (Participants) | 10
kPa
  Month 12: number analyzed (Participants) | 6
  Month 12 | -1.15 [-9.60 to 0.40]
  Month 24/EOT: number analyzed (Participants) | 6
  Month 24/EOT | -1.70 [-4.20 to -0.90]

47. Secondary Outcome: Median Change From Baseline In Total Bile Acids
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24/EOT
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: umol/L
Arm/Group | Long-term Safety Extension Phase
Number analyzed (Participants) | 20
umol/L
  Month 6: number analyzed (Participants) | 19
  Month 6 | -1.56 [-5.23 to 2.58]
  Month 12: number analyzed (Participants) | 19
  Month 12 | -1.14 [-8.94 to 2.88]
  Month 18: number analyzed (Participants) | 17
  Month 18 | -4.61 [-9.21 to 2.80]
  Month 24/EOT: number analyzed (Participants) | 17
  Month 24/EOT | -4.91 [-9.81 to 1.10]

48. Secondary Outcome: Median Change From Baseline In Total Endogenous Bile Acid
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24/EOT
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: umol/L
Arm/Group | Long-term Safety Extension Phase
Number analyzed (Participants) | 20
umol/L
  Month 6: number analyzed (Participants) | 19
  Month 6 | -0.83 [-3.17 to -0.09]
  Month 12: number analyzed (Participants) | 19
  Month 12 | -0.77 [-3.54 to 0.18]
  Month 18: number analyzed (Participants) | 17
  Month 18 | -2.19 [-4.62 to -0.48]
  Month 24/EOT: number analyzed (Participants) | 17
  Month 24/EOT | -2.02 [-4.22 to 0.98]

49. Secondary Outcome: Median Change From Baseline In Total UDCA
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24/EOT
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: umol/L
Arm/Group | Long-term Safety Extension Phase
Number analyzed (Participants) | 20
umol/L
  Month 6: number analyzed (Participants) | 19
  Month 6 | -0.34 [-2.67 to 3.47]
  Month 12: number analyzed (Participants) | 19
  Month 12 | -0.47 [-4.19 to 2.69]
  Month 18: number analyzed (Participants) | 17
  Month 18 | -2.89 [-4.95 to 2.50]
  Month 24/EOT: number analyzed (Participants) | 17
  Month 24/EOT | -1.68 [-6.17 to 0.50]

50. Secondary Outcome: Median Change From Baseline In Total Chenodeoxycholic Acid
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24/EOT
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: umol/L
Arm/Group | Long-term Safety Extension Phase
Number analyzed (Participants) | 20
umol/L
  Month 6: number analyzed (Participants) | 19
  Month 6 | -0.20 [-0.85 to 0.07]
  Month 12: number analyzed (Participants) | 19
  Month 12 | -0.35 [-1.69 to 0.10]
  Month 18: number analyzed (Participants) | 17
  Month 18 | -1.28 [-1.84 to -0.06]
  Month 24/EOT: number analyzed (Participants) | 17
  Month 24/EOT | -1.17 [-1.76 to 0.33]

51. Secondary Outcome: Median Change From Baseline In Total Lithocholic Acid
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24/EOT
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: umol/L
Arm/Group | Long-term Safety Extension Phase
Number analyzed (Participants) | 20
umol/L
  Month 6: number analyzed (Participants) | 19
  Month 6 | 0.00 [-0.03 to 0.11]
  Month 12: number analyzed (Participants) | 19
  Month 12 | 0.00 [-0.05 to 0.06]
  Month 18: number analyzed (Participants) | 17
  Month 18 | 0.00 [-0.10 to 0.00]
  Month 24/EOT: number analyzed (Participants) | 17
  Month 24/EOT | 0.00 [-0.19 to 0.00]

52. Secondary Outcome: Median Change From Baseline In Total Cholic Acid
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24/EOT
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: umol/L
Arm/Group | Long-term Safety Extension Phase
Number analyzed (Participants) | 20
umol/L
  Month 6: number analyzed (Participants) | 19
  Month 6 | -0.39 [-1.39 to 0.00]
  Month 12: number analyzed (Participants) | 19
  Month 12 | -0.48 [-1.44 to 0.00]
  Month 18: number analyzed (Participants) | 17
  Month 18 | -0.49 [-1.49 to -0.09]
  Month 24/EOT: number analyzed (Participants) | 17
  Month 24/EOT | -0.39 [-1.18 to -0.04]

53. Secondary Outcome: Median Change From Baseline In Total Deoxycholic Acid
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24/EOT
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: umol/L
Arm/Group | Long-term Safety Extension Phase
Number analyzed (Participants) | 20
umol/L
  Month 6: number analyzed (Participants) | 19
  Month 6 | -0.59 [-0.89 to -0.04]
  Month 12: number analyzed (Participants) | 19
  Month 12 | -0.56 [-1.14 to 0.01]
  Month 18: number analyzed (Participants) | 17
  Month 18 | -0.51 [-1.21 to -0.27]
  Month 24/EOT: number analyzed (Participants) | 17
  Month 24/EOT | -0.59 [-1.10 to 0.32]

54. Secondary Outcome: Absolute Change From Baseline In HDL Cholesterol Concentration
Time Frame: Baseline, Month 24/EOT
Population: as for outcome 46
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Long-term Safety Extension Phase
Number analyzed (Participants) | 17
mmol/L | 0.5 [-4.6 to 5.5]
Statistical Analysis 1: Comparison: Long-term Safety Extension Phase; Test type: Superiority or Other; p = 0.852, ANCOVA

55. Secondary Outcome: Absolute Change From Baseline In HDL Particle Size
Time Frame: Baseline, Month 24/EOT
Population: as for outcome 46
Measure: Least Squares Mean (95% Confidence Interval); unit: nm
Arm/Group | Long-term Safety Extension Phase
Number analyzed (Participants) | 17
nm | 0.04 [-0.10 to 0.19]
Statistical Analysis 1: Comparison: Long-term Safety Extension Phase; Test type: Superiority or Other; p = 0.549, ANCOVA

56. Secondary Outcome: Absolute Change From Baseline In HDL Particle Number
Time Frame: Baseline, Month 24/EOT
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: umol/L
Arm/Group | Long-term Safety Extension Phase
Number analyzed (Participants) | 20
umol/L | -0.09 [-1.78 to 1.59]
Statistical Analysis 1: Comparison: Long-term Safety Extension Phase; Test type: Superiority or Other; p = 0.912, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of the first dose of investigational product until the participant fully completed participation in the study, up to 2 years.
Arm/Group | Primary Treatment Phase | Long-term Safety Extension Phase
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/21
Serious Adverse Events (participants affected / at risk) | 1/26 | 5/21
Other Adverse Events (participants affected / at risk) | 18/26 | 17/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Treatment Phase (N=26) | Long-term Safety Extension Phase (N=21)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Treatment Phase (N=26) | Long-term Safety Extension Phase (N=21)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (17) | 6 (13)
Fatigue (General disorders) | 4 (4) | 0 (0)
Oedema peripheral (General disorders) | 2 (3) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (4) | 2 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2)
Low density lipoprotein increased (Investigations) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Tooth abscess (Infections and infestations) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dry eye (Eye disorders) | 0 (0) | 2 (2)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators must wait 18 months after the study ends to publish their results and a multi-center publication must come first. The sponsor has a 45 day review period with the option to extend to an additional 90 days.